CLINICAL TRIAL: NCT02716415
Title: Randomized Controlled Trial Comparing the Efficacy and Safety of Calmoseptine Ointment and Desitin Maximum Strength 40% Zinc Oxide Diaper Rash Paste in Diaper Dermatitis in Neonates and Infants
Brief Title: Trial Comparing Calmoseptine Ointment and Desitin Diaper Rash Paste in Diaper Dermatitis in Neonates and Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of the Philippines (Other)
Collaborators: Calmoseptine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-019-01
Record Dates: First submitted 2016-02-24; First posted 2016-03-23 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Diaper Dermatitis
Keywords: neonates; infants
MeSH Terms: conditions — Diaper Rash | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calmoseptine Ointment (Active Comparator): Calmoseptine Ointment as part of a structured skin care regimen.
  Interventions: Drug: Calmoseptine Ointment
- Destin Maximum Strength 40% Zinc (Active Comparator): Destin Maximum Strength 40% Zinc as part of a structured skin care regimen.
  Interventions: Drug: Destin Maximum Strength 40% Zinc

INTERVENTIONS:
Drug: Calmoseptine Ointment — A full structured skin care regimen is provided in a consistent fashion either by study personnel or by the participant's primary carer (family or ward staff) at each diaper change. Study nurse sub-investigator visit each participant twice per nursing shift (six times per day) either to deliver the care regimen or to observe that it is being delivered.
  The regimen includes:
  * regular diaper changing,
  * gentle cleansing
  * application of the trial ointment
  Other Names: Calmoseptine
  Arms: Calmoseptine Ointment
Drug: Destin Maximum Strength 40% Zinc — A full structured skin care regimen is provided in a consistent fashion either by study personnel or by the participant's primary carer (family or ward staff) at each diaper change. Study nurse sub-investigator visit each participant twice per nursing shift (six times per day) either to deliver the care regimen or to observe that it is being delivered.
  The regimen includes:
  * regular diaper changing,
  * gentle cleansing
  * application of the trial ointment
  Other Names: Destin
  Arms: Destin Maximum Strength 40% Zinc

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Calmoseptine Ointment and Desitin Maximum Strength 40% Zinc Oxide Diaper Rash Paste in the treatment of diaper dermatitis among Neonates and Infants.

DETAILED DESCRIPTION:
This is a single-center, randomized, controlled, assessor-blinded clinical trial. Neonates born in UP-PGH or infants (< 1 year of age) in the general pediatric wards for any condition who have diaper dermatitis are recruited and randomized to treatment with either Calmoseptine Ointment or Desitin Maximum Strength 40% Zinc Oxide Diaper Rash Paste as part of a structured skin care regimen. Each participant has one week total participation, unless withdrawn. Baseline data are collected and study treatment initiated on study entry day. Treatment continued and follow up data collected on six subsequent follow up days. Primary outcome: healing of Diaper Dermatitis after six days of treatment, defined as a Diaper Dermatitis Severity Score of zero attributed by blinded assessment. Secondary outcomes: Diaper Dermatitis Severity Score at each day of treatment; size of affected area; incidence of Candida infection; adverse events.

Zinc Oxide Ointment preparations including Calmoseptine Ointment and Desitin Maximum Strength 40% Diaper Rash Paste have been used to treat diaper dermatitis for many years around the world. There are no known reported hypersensitivities to either product and no reported serious adverse events. As the proposed study is in neonates and infants, as a precaution the evidence relating to the safety and toxicity of individual ingredients were reviewed for the trial protocol prior to commencement.

ELIGIBILITY:
Inclusion Criteria:

1. The child participant must be < 1 year of age.
2. The participant must, upon clinical inspection by an investigator, be assessed to have diaper dermatitis ≥ Grade 2 according to the study's diaper dermatitis severity scale (see "Primary Outcome").
3. The participant's parent, next of kin or legally acceptable representative agrees to the child's inclusion and signs the informed consent.
4. The participant's primary physician agrees to inclusion.
5. There is a reasonable expectation that the participant will be hospitalized for at least 7 days and will be able to complete the study. (NB Study Participant Withdrawal Criteria b - Any participants discharged from hospital by their attending physician before completion of study participation will automatically be withdrawn from the study. Study participation will not under any circumstances lead to delay in a participant's discharge from hospital.)
6. Participant has no known allergy or history of adverse reaction to any of the ingredients in either product or to any topical preparations or skin care products

Exclusion Criteria:

1. Participants with a pre-existing full thickness wound within the study area.
2. Participants with pre-existing active dermatological condition(s), other than DD, which may affect healing or interpretation of trial results. Where uncertainty exists, the Investigators will arrange a consultation with a Consultant Dermatologist.
3. Participant has a history of recurrent dermatological conditions, other than DD, that may imply difficult healing or affect interpretation of trial results.
4. Participant has any severe acute or chronic medical condition such that trial participation may constitute a risk, or may interfere with their medical care, or affect interpretation of results, or their attending physician advises against participation.
5. Participant is on systemic antifungal treatment (eg. Amphotericin B or Fluconazole), topical antifungal treatment and / or systemic or topical corticosteroids.
6. Participant has in the preceding week been treated with topical agents that may affect healing (e.g. dimethicone based ointments, zinc oxide powder, petroleum jelly)

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 319 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Healing of diaper Dermatitis | Assessed on Final day of data collection (Day 6)
  Complete healing of Diaper Dermatitis on final study day, as determined by Diaper Dermatitis Severity Scale. Possible score range from zero (0 - clear skin) ti six (6 - severe erythema, all or most of the diaper area affected, with papules and/or pustules, and open skin affecting the dermis). Complete healing is defined as a Diaper Dermatitis Severity Score of zero (0).
  Assessment of the primary outcome used in final analyses will be blinded. For determination of final trial results for the primary outcome, sets of high definition photographs for each patient on each treatment day will be assessed by independent wound, Ostomy and Continence Nursing Certification Board (WOCNB) certified wound care expert assessors based in the USA, who are blinded to treatment allocation, not involved in the study.

SECONDARY OUTCOMES:
Daily Diaper Dermatitis Severity Score | Assessed on Day 0, 1, 2, 3, 4, 5, and 6
  Diaper dermatitis severity, assessed as per primary outcome.
  The size of area affected by diaper dermatitis is measured and recorded at baseline (study entry on Day 0) and on each follow up day (Days 1-6). Disposable paper tape measures are used to prevent cross-infection. Where more than one non-contiguous area is affected, each will be measured as described and added together. As the study will include neonates and infants up to one year of age, body size will differ significantly so that an affected area of a similar size may be more serious in one participant than in another. Accordingly, the mean body size and/or weight of treatment groups will be considered and the expression of area affected used in final analyses will be adjusted appropriately.

OTHER OUTCOMES:
Size of area affected by diaper dermatitis on Days 0-6. | Measured on Day 0, 1, 2, 3, 4, 5, and 6
  The area will be calculated by multiplying the longest portion of the affected area measured in a head to toe orientation by the widest portion of the affected area measured from side to side (in centimeters).
Adverse Events. | Recorder on Day 0, 1, 2, 3, 4, 5, and 6
  Non-Serious and serious adverse events judged by physicians to be due to trial participation.

CONTACTS AND LOCATIONS:
Overall Officials: Jacinto Blas Mantaring, MD, Principal Investigator — Department of Pediatrics, Philippine General Hospital UP Manila
Locations (1):
- Philippine General Hospital - University of the Philippines, Manila, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No